CLINICAL TRIAL: NCT01281488
Title: A Prospective Investigation of the Use of the Fluorescence Imaging on the da Vinci Surgical System for Intraoperative Near Infrared Imaging of Renal Cortical Tumors
Brief Title: Fluorescence Imaging in Finding Tumors in Patients With Kidney Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 10155; NCI-2011-00067 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-01-19; First posted 2011-01-24 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Recurrent Renal Cell Cancer; Stage I Renal Cell Cancer; Stage II Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Optical Imaging; Laparoscopy; Indocyanine Green

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Treatment 1 (fluorescence imaging and surgery) (Experimental): Patients undergo NIR fluorescence imaging with ICG and an additional 0.018 mg/kg/dose on the da Vinci Surgical System followed by standard approach robot-assisted laparoscopic partial nephrectomy.
  Interventions: Procedure: fluorescence imaging; Procedure: laparoscopic surgery; Drug: indocyanine green
- Treatment 2 (fluorescence imaging and surgery) (Experimental): Patients undergo NIR fluorescence imaging with ICG and an additional 0.036 mg/kg/dose on the da Vinci Surgical System followed by standard approach robot-assisted laparoscopic partial nephrectomy.
  Interventions: Procedure: fluorescence imaging; Procedure: laparoscopic surgery; Drug: indocyanine green
- Treatment 3 (fluorescence imaging and surgery) (Experimental): Patients undergo NIR fluorescence imaging with ICG and an additional 0.07 mg/kg/dose on the da Vinci Surgical System followed by standard approach robot-assisted laparoscopic partial nephrectomy.
  Interventions: Procedure: fluorescence imaging; Procedure: laparoscopic surgery; Drug: indocyanine green
- Treatment 4 (fluorescence imaging and surgery) (Experimental): Patients undergo NIR fluorescence imaging with ICG and an additional 0.14 mg/kg/dose on the da Vinci Surgical System followed by standard approach robot-assisted laparoscopic partial nephrectomy.
  Interventions: Procedure: fluorescence imaging; Procedure: laparoscopic surgery; Drug: indocyanine green
- Treatment 5 (fluorescence imaging and surgery) (Experimental): Patients undergo NIR fluorescence imaging with ICG and an additional 0.21 mg/kg/dose on the da Vinci Surgical System followed by standard approach robot-assisted laparoscopic partial nephrectomy.
  Interventions: Procedure: fluorescence imaging; Procedure: laparoscopic surgery; Drug: indocyanine green

INTERVENTIONS:
Procedure: fluorescence imaging — Undergo NIR fluorescence imaging with ICG on the da Vinci surgical system
Procedure: laparoscopic surgery — Undergo standard approach robot-assisted laparoscopic partial nephrectomy
  Other Names: laparoscopy-assisted surgery; surgery, laparoscopic
Drug: indocyanine green — Given IV

SUMMARY:
RATIONALE: Using fluorescence imaging may determine the extent of kidney tumors and help in planning surgery.

PURPOSE: This phase I trial is studying the best way to give indocyanine green (ICG) fluorescence imaging in finding tumors in patients with kidney tumors

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the optimal dose of ICG fluorescence for visualization using the SPY scope with near infrared (NIR) imaging technology on the da Vinci Surgical System to detect renal cortical tumors and to assist in their removal.

SECONDARY OBJECTIVES:

I. To observe and report peri-operative outcomes, including but not limited to the following observations: positive surgical margin rate, correlation of the ICG and NIR imaging technology with intraoperative ultrasound imaging and preoperative imaging, incidence of adverse events, estimated blood loss, blood transfusion rate, length of stay, time of operation, utility of ICG and NIR imaging technology to assist in localization of renal hilar structures, utility of ICG and NIR imaging technology to assist in localization of the renal mass, warm renal ischemia time measurements, the feasibility of selective renal arterial clamping with the ICG and NIR imaging technology, cost analysis retrospective comparisons to patients who underwent similar surgical procedures without the use of ICG and NIR imaging technology, the overall effect of ICG and NIR imaging technology on postoperative renal function, and determination of possible future technique variations using the ICG and NIR imaging technology to improve nephron sparing surgery.

OUTLINE: This is a dose-escalation study. Patients undergo NIR fluorescence imaging with ICG on the da Vinci Surgical System followed by standard approach robot-assisted laparoscopic partial nephrectomy.

After completion of study treatment, patients are followed up at 1-2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a computed tomography (CT) scan or magnetic resonance imaging (MRI) on preoperative assessment showing evidence of a renal cortical tumor; the renal tumor must be stage T1a/bT2
* Due to concerns of surgical and anesthetic effects on the fetus, women of child bearing age who are considered to still be fertile must undergo a urine pregnancy test prior to inclusion in the study; only women with negative urine pregnancy tests prior to surgery will be included; if a women is found to have a positive urine pregnancy test, surgery and potential inclusion in the study will be deferred until after delivery of the baby; should a woman become pregnant or suspect that she is pregnant prior to surgical management, she should inform her treating physician immediately; although it is known that ICG is released from the body through the hepatic system, breastfeeding mothers will be excluded from the study due to the unknown side effects on the infant in the breastfeeding population
* The subject must be able to comply with the study procedures
* All subjects must have the ability to understand the risks, benefits, and alternatives of the study and the willingness to sign a written informed consent

Exclusion Criteria:

* Subject has significant liver disease, cirrhosis or liver insufficiency with abnormal liver function tests, as total bilirubin greater than 1.5 X normal and/or serum glutamic oxaloacetic transaminase (SGOT) greater than 2 X normal
* Subject has uremia, serum creatinine greater than 2.0 mg/dl
* Subject has previous history of adverse reaction or allergy to ICG, iodine, shellfish or iodine dyes
* Subject in whom the use of x ray dye or ICG is contraindicated including development of adverse events when previously or presently administered
* Subject has any medical condition, which in the judgment of the Investigator and/or designee makes the subject a poor candidate for the investigational procedure
* Subject is actively participating in another drug, biologic and/or device protocol
* The presence of medical conditions contraindicating general anesthesia or standard surgical approaches
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-10-20; Primary Completion 2017-10-09 (Actual); Study Completion 2017-10-09 (Actual)

PRIMARY OUTCOMES:
Determination of the optimal dose of ICG which will maximize its utility in the detection of renal cortical tumors by NIR imaging technology on the da Vinci Surgical System | 2 weeks post surgery
  Compared between patients prospectively accrued to the study who had fluorescence imaging and those in the retrospective cohort whose procedures were not assisted with fluorescence imaging.

SECONDARY OUTCOMES:
Positive margin from pathology | 2 weeks post-surgery
  Compared between patients prospectively accrued to the study who had fluorescence imaging and those in the retrospective cohort whose procedures were not assisted with fluorescence imaging.
Total surgical time | At surgery
  Compared between patients prospectively accrued to the study who had fluorescence imaging and those in the retrospective cohort whose procedures were not assisted with fluorescence imaging.
Warm ischemia time | At surgery
  Compared between patients prospectively accrued to the study who had fluorescence imaging and those in the retrospective cohort whose procedures were not assisted with fluorescence imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Lau, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States